CLINICAL TRIAL: NCT05222828
Title: Evaluation of the Efficacy and Safety of Mepivacaine on the Neurological Sequelae of Cerebral Infarction
Brief Title: Effects of Mepivacaine on the Neurological Sequelae of Cerebral Infarction
Acronym: MEPI-AVC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190723; 2021-005507-13 (EudraCT Number)
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mepivacaine arm (Experimental): mepivacaine injection
  Interventions: Drug: Carbocaine Injectable Product

INTERVENTIONS:
Drug: Carbocaine Injectable Product — One injection per patient

SUMMARY:
A patient, suffering from cortical blindness after a bi-occipital infarction 1 year earlier, regained near-normal vision in the right visual hemifield a few minutes after subcutaneous administration of mepivacaine. The effect was maintained for several days, and was repeated with each injection of mepivacaine. This clinical improvement is associated with functional changes in the peri-lesional areas on resting-state functional MRI.

The investigator team hypothesizes that in some patients with chronic neurological symptoms of stroke, the investigator team will observe a favorable response to subcutaneous mepivacaine injection.

DETAILED DESCRIPTION:
A patient, suffering from cortical blindness after a bi-occipital infarction 1 year earlier, regained near-normal vision in the right visual hemifield a few minutes after subcutaneous administration of mepivacaine. The effect was maintained for several days, and was repeated with each injection of mepivacaine. This clinical improvement is associated with functional changes in the peri-lesional areas on resting-state functional MRI. The investigator team hypothesizes that in some patients with chronic neurological symptoms of stroke, investigator team will observe a favorable response to subcutaneous mepivacaine injection.

The team will include patients with clinically significant sequelae of ischemic stroke, as was the case with the initial patient. In addition,

* The team hypothesizes that the mechanism of action is not specific to the visual cortex, and therefore should not be limited to visual scotomas
* It is also preferable to consider only deficits that can be objectively quantified in a sufficiently reliable way to be able to evaluate the effect of the treatment

The investigator teamwill therefore include patients with sequelae of at least one of the following three types:

* motor deficit: score =< 56 on the Fugl-Meyer scale, minimal deficit allowing to observe an improvement of 4 points
* aphasia: score >= 4 on the Aphasia Rapid Test (ART) , minimal deficit allowing to observe an improvement of 4 points
* visual scotoma: observable on a clinical assessment of the visual field "on confrontation"

Only patients more than 30 days after the occurrence of the stroke will be included. Indeed, the rapid recovery phase after a stroke lasts about 3 weeks and it is difficult to interpret rapid clinical changes and to attribute them to the treatment (since investigator team do not know the time of onset of the effect of mepivacaine) over this temporal period.

Mepivacaine will be administered as a single injection, subcutaneously, at a dose of 3 mL of mepivacaine hydrochloride (20 mg/mL), or 60mg. If mepivacaine is effective, research participants will experience a temporary reduction in neurological symptoms.

Time course of experiment

1. Signing of consent
2. Verification of inclusion and exclusion criteria (1h)

   * ECG for all patients
   * Urine dipstick if female of childbearing age
   * Motor, language and visual field scales, depending on the deficit(s) present
3. Blood sampling
4. Evaluation of the neurological deficit before treatment (1h)

   * VAS to evaluate the intensity of symptoms by the patient
   * NIHSS
5. MRI n°1 (duration 45 min to 1h)
6. Administration of mepivacaine 7 Evaluation of the neurological deficit after treatment, at T= 1+/- 30 minutes after administration (duration 1h)

   * Motor, language and visual field scales, depending on the deficit(s) present
   * VAS to evaluate the intensity of the symptoms by the patient
   * NIHSS

8/ MRI n°2 (duration 30 to 45min) 1h30 after administration 9/ Evaluation of the neurological deficit after treatment, at T= 3h45+/- 45 minutes after administration (duration 1h)

* Motor, language and visual field scales, depending on the deficit(s) present
* VAS to evaluate the intensity of the symptoms by the patient
* NIHSS 9/ Call of the patient 1 week later for follow-up of SAEs and evaluation of the duration of the effect, if any ; if the effect persists, the investigator will call the patient every 2 weeks until returning to the usual state..

Brain imaging

MRI will be performed on a SIEMENS 3 Tesla machine, without injection of contrast medium. The duration of the MRI will be approximately 45 minutes to one hour for MRI n°1 (baseline) and 30 to 45 minutes for MRI n°2 performed after the injection of mepivacaine.

MRI acquisitions will include the following sequences:

* T1 (only during MRI n°1 in baseline)
* FLAIR (only during baseline MRI n°1)
* Diffusion sequence (multishell, multiband)
* Perfusion sequence (Arterial Spin Labelling, ASL)
* Resting state BOLD sequence

Drug treatment :

Mepivacaine will be administered:

* Subcutaneously
* In the shoulder on the non-dominant side, or on the non-deficient side in case of hemiplegia
* Dose: 3 mL of mepivacaine hydrochloride (20 mg/mL), or 60mg
* With at disposal

  * Resuscitation equipment (in particular, a source of oxygen)
  * lipid emulsion to be administered in case of intoxication with clinical signs of neurotoxicity or cardiotoxicity

Genetic samples :

The gene coding for brain-derived neurotrophic factor (BDNF) is of particular interest. BDNF is a protein that contributes to neurogenesis and neuronal differentiation, participates in the creation of new synapses and influences the survival of existing neurons. It is thus currently considered as a crucial element influencing brain plasticity . This could also be an explanatory factor in identifying responders to mepivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke more than 30 days old
* Age between 18 and 85 years old
* At least one deficit among:
* motor deficit: score < 56 on the Fugl-Meyer scale
* aphasia: score ≥4 on the Aphasia Rapid Test,
* presence of a clinically observable visual scotoma
* Having given their written consent
* Be affiliated with a social security scheme, Universal Medical Coverage (CMU) or any equivalent scheme

Exclusion Criteria:

* Hypersensitivity to amide-bonded local anesthetics.
* Atrioventricular conduction disorders requiring permanent electro-systolic training not yet performed.
* Epilepsy not controlled by treatment.
* Porphyritic subjects.
* Patients with a motor deficit (but no aphasia or scotomas) in whom there is spasticity leading to a major reduction in joint amplitude in passive motion
* Minor patients, under curatorship or guardianship, under legal protection, deprived of liberty, pregnant or breastfeeding women
* Pathologies involving the vital prognosis or compromising follow-up during the study period
* Patient undergoing local amine anesthesia in the 7 days preceding V1.
* Patients currently treated with no anti-arrhythmics such as tocainide, aprindine and mexiletine
* Patients with a contraindication to MRI (ferro-magnetic surgical clips, eye implants, metallic foreign body intraocular or in the nervous system, implants or metallic objects likely to contain the radiofrequency field, cochlear implants, cerebral or cardiac pacemaker , implantable cardiac defibrillators)
* Patients participating in research involving the therapeutic human person who may modify functional recovery (whether by medication or by medical device) or subject to an exclusion period for another research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
improvement of clinical scores | 1 Day
  The response is defined as an improvement 1h (+/- 30min) after injection, compared to the evaluation before mepivacaine injection, on at least one of the clinical scores specific to the symptoms:
  * language : decrease of at least 4 points on the ART scale (rated from 0 to 26) , or increase of 20% of the number of images correctly named on a standardized battery (DO80, rated from 0 to 80). The rate of 20% corresponds to an effect considered clinically significant, without any "clinically significant minimal change" published to date.
  * motor skills : increase of at least 4 points on the Fugl-Meyer scale (rated from 0 to 60) corresponding to the "clinically significant minimal change" in the re-education studies
  * visual field : 20% reduction of a scotoma evaluated in automated static perimetry of Humphrey by the number of deficit areas compared to the total number of areas evaluated (n=43). The rate of 20% corresponds to an effect considered clinically significant

SECONDARY OUTCOMES:
language-related symptoms | 1 Day
  Relative change, in percentage, in the number of correctly named images on a standardized battery (DO80, rated from 0 to 80) between pre- and 1h(+/-30min) post-injection to measure language-related symptoms.
ART scale | 1 Day
  Absolute change, in number of points, on the ART scale (rated from 0 to 26) between before and 1h(+/-30min) after injection to measure language-related symptoms.
spontaneous language test | 1 Day
  Relative change, of he rate from 0 to 10 at the spontaneous language test between before and 1h(+/-30min) after injection to measure language-related symptoms.
Fugl-Meyer scale | 1Day
  Absolute change, in number of points, on the Fugl-Meyer scale (rated from 0 to 60), between before and 1h(+/-30min) after injection to measure motor symptoms.
Timed up and go test | 1Day
  relative change, on the Timed up and go test (TUG) (rated in seconds), between before and 1h(+/-30min) after injection to measure motor symptoms.
10 metres walking test | 1Day
  Relative change, on the 10 metres walking test (rated in seconds), between before and 1h(+/-30min) after injection to measure motor symptoms.
Perimetry of Humphrey | 1 Day
  Relative evolution of visual symptoms, measured in automated static perimetry of Humphrey (STAT-30, Metrovision) by the number of deficit areas compared to the total number of assessed areas (n=43), between before and 1h (+/-30min) after injection
kinetic perimetry | 1 Day
  Relative evolution of visual symptoms, measured in kinetic perimetry by the surface of isoptera III/4, between before and 1h (+/-30min) after injection.
static perimetry | 1 Day
  Evolution of visual deficit volumes, measured in static perimetry in dB.deg2, between before and 1h (+/-30min) after injection.
NIHSS score changes | 1 Day
  Change in severity of neurological sequelae measured by the relative change in the National Institutes of Health Stroke Scale (NIHSS score) between before and 1h(+/-30min) after injection.
response delay | 1 Day
  Patient Reported Response Start and End Times

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpetrière, Paris, France